CLINICAL TRIAL: NCT01008371
Title: CCK-dysregulation: Mechanisms of Abnormal Food Regulation and Obesity
Brief Title: Investigation of Neuro-hormonal Mechanisms of Hunger, Fullness and Obesity.
Status: Withdrawn | Type: Observational
Why Stopped: No recruitment
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Society of Nuclear Medicine (Unknown)
Responsible Party: Kelly Holes-Lewis, M.D., Medical University of South Carolina
Other Study IDs: 19449
Record Dates: First submitted 2009-11-03; First posted 2009-11-05 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2010-07

CONDITIONS: Obesity; Gastric Emptying; Anxiety; Depression; Panic Disorder
Keywords: Obesity; Cholecystokinin; Oxytocin; Satiety; Gastric emptying; Anxiety; Depression; Panic Disorder
MeSH Terms: conditions — Obesity; Anxiety Disorders; Depression; Panic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese: Healthy obese subjects
- Non-obese: Healthy non-obese subjects

SUMMARY:
The purpose of this study is to determine abnormal neuro-hormonal mechanisms that may impair the ability to feel full and which therefore, may lead to obesity.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 to 65 years of age.
* Obese Subjects with BMI >40.
* Normal weight subjects with BMI = 18.5-24.9

Exclusion Criteria:

* Age younger than 18 years and over 65 years of age.
* Current use of narcotics or morphine
* Previous gastric surgery
* Presence of the following disorders that are known to cause functional gastric stasis syndromes: Diabetes Mellitus, Hypothyroidism, Progressive Systemic Sclerosis, Systemic Lupus Erythematosus, Dermatomyositis, Familial Dysautonomia, Pernicious Anemia, Bulbar poliomyelitis, Amyloidosis, Gastric Ulcer, Post-vagotomy, Tumor-associated gastroparesis, Fabry disease, Myotonic Dystrophy, Post-operative ileus, Gastroenteritis.
* Presence of the following disorders that are known to cause delayed gastric emptying: peptic ulceration, recent surgery, pyloric hypertrophy, post-radiotherapy, ileus, anorexia nervosa, acute viral infections.
* Presence of the following disorders that are known to cause rapid gastric emptying: Pyloroplasty, Hemigastrectomy, Duodenal ulcer, Gastrinoma (Zollinger-Ellison syndrome), Hyperthyroidism
* Current use of Thyroxine as it is known to cause rapid gastric emptying
* Current or recent (within the last 2 weeks) use of anti-spasmodics or pro-kinetic medications.
* Current use of Hyperalimentation
* Presence of any metabolic disorder, such as: hyperglycemia, acidosis, hypokalemia, hypercalcemia, hepatic coma or myxedema.
* Current use of estrogen or progesterone
* Current use of the following drugs that are known to delay gastric emptying: Nifedipine, beta-adrenergic agonists, Isoproterenol, Theophylline, Sucralfate, anticholinergics, Levodopa, diazepam, tricyclic antidepressants, phenothiazine, Progesterone, oral contraceptives, alcohol, nicotine, opiates.
* Allergy to eggs or wheat.
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample, patients of a weight management clinic and patients of Medical University of South Carolina
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Cholecystokinin serum level | fasting- state, then at time points 30, 60 and 120 minutes post-meal
Oxytocin serum bioassay | fasting-state, and then at time points of 30, 60 and 120 minutes post-meal
Gastric Emptying time | calculated at time points 0.5, 1,2,3 and 4 hours post-meal
Perception of fullness using visual analog scales | fasting-state, and then at time points of every half hour post-meal through completion of the scan

SECONDARY OUTCOMES:
Mini International Neuro-psychiatric Interview (MINI) | once within 30 days of the scan

CONTACTS AND LOCATIONS:
Overall Officials: Kelly A Holes-Lewis, M.D., Principal Investigator — Medical University of South Carolina; Thomas W Uhde, M.D., Study Chair — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Flegal KM, Graubard BI, Williamson DF, Gail MH. Cause-specific excess deaths associated with underweight, overweight, and obesity. JAMA. 2007 Nov 7;298(17):2028-37. doi: 10.1001/jama.298.17.2028. PMID 17986696
- [Background] Clinical guidelines on the identification, evaluation, and treatment of overweight and obesity in adults: executive summary. Expert Panel on the Identification, Evaluation, and Treatment of Overweight in Adults. Am J Clin Nutr. 1998 Oct;68(4):899-917. doi: 10.1093/ajcn/68.4.899. No abstract available. PMID 9771869
- [Background] Valassi E, Scacchi M, Cavagnini F. Neuroendocrine control of food intake. Nutr Metab Cardiovasc Dis. 2008 Feb;18(2):158-68. doi: 10.1016/j.numecd.2007.06.004. Epub 2007 Dec 3. PMID 18061414
- [Background] Burton-Freeman B, Davis PA, Schneeman BO. Plasma cholecystokinin is associated with subjective measures of satiety in women. Am J Clin Nutr. 2002 Sep;76(3):659-67. doi: 10.1093/ajcn/76.3.659. PMID 12198015
- [Background] Konturek SJ, Konturek JW, Pawlik T, Brzozowski T. Brain-gut axis and its role in the control of food intake. J Physiol Pharmacol. 2004 Mar;55(1 Pt 2):137-54. PMID 15082874
- [Background] Rehfeld JF. Accurate measurement of cholecystokinin in plasma. Clin Chem. 1998 May;44(5):991-1001. PMID 9590372
- [Background] Liddle RA, Morita ET, Conrad CK, Williams JA. Regulation of gastric emptying in humans by cholecystokinin. J Clin Invest. 1986 Mar;77(3):992-6. doi: 10.1172/JCI112401. PMID 3949984
- [Background] McCann UD, Slate SO, Geraci M, Roscow-Terrill D, Uhde TW. A comparison of the effects of intravenous pentagastrin on patients with social phobia, panic disorder and healthy controls. Neuropsychopharmacology. 1997 Mar;16(3):229-37. doi: 10.1016/S0893-133X(96)00197-2. PMID 9138439
- [Background] Zhang W, Gardell S, Zhang D, Xie JY, Agnes RS, Badghisi H, Hruby VJ, Rance N, Ossipov MH, Vanderah TW, Porreca F, Lai J. Neuropathic pain is maintained by brainstem neurons co-expressing opioid and cholecystokinin receptors. Brain. 2009 Mar;132(Pt 3):778-87. doi: 10.1093/brain/awn330. Epub 2008 Dec 2. PMID 19050032
- [Background] Moran TH, Dailey MJ. Minireview: Gut peptides: targets for antiobesity drug development? Endocrinology. 2009 Jun;150(6):2526-30. doi: 10.1210/en.2009-0003. Epub 2009 Apr 16. PMID 19372201
- [Background] Konturek PC, Konturek JW, Czesnikiewicz-Guzik M, Brzozowski T, Sito E, Konturek SJ. Neuro-hormonal control of food intake: basic mechanisms and clinical implications. J Physiol Pharmacol. 2005 Dec;56 Suppl 6:5-25. PMID 16340035
- [Background] Little TJ, Russo A, Meyer JH, Horowitz M, Smyth DR, Bellon M, Wishart JM, Jones KL, Feinle-Bisset C. Free fatty acids have more potent effects on gastric emptying, gut hormones, and appetite than triacylglycerides. Gastroenterology. 2007 Oct;133(4):1124-31. doi: 10.1053/j.gastro.2007.06.060. Epub 2007 Jul 3. PMID 17919488
- [Background] Monstein HJ, Grahn N, Truedsson M, Ohlsson B. Oxytocin and oxytocin-receptor mRNA expression in the human gastrointestinal tract: a polymerase chain reaction study. Regul Pept. 2004 Jun 15;119(1-2):39-44. doi: 10.1016/j.regpep.2003.12.017. PMID 15093695
- [Background] Ohlsson B, Forsling ML, Rehfeld JF, Sjolund K. Cholecystokinin stimulation leads to increased oxytocin secretion in women. Eur J Surg. 2002;168(2):114-8. doi: 10.1080/11024150252884340. PMID 12113268
- [Background] Borg J, Melander O, Johansson L, Uvnas-Moberg K, Rehfeld JF, Ohlsson B. Gastroparesis is associated with oxytocin deficiency, oesophageal dysmotility with hyperCCKemia, and autonomic neuropathy with hypergastrinemia. BMC Gastroenterol. 2009 Feb 25;9:17. doi: 10.1186/1471-230X-9-17. PMID 19243587
- [Background] Runge CF. Economic consequences of the obese. Diabetes. 2007 Nov;56(11):2668-72. doi: 10.2337/db07-0633. Epub 2007 Jun 29. PMID 17601989
- [Background] Dall TM, Fulgoni VL 3rd, Zhang Y, Reimers KJ, Packard PT, Astwood JD. Potential health benefits and medical cost savings from calorie, sodium, and saturated fat reductions in the American diet. Am J Health Promot. 2009 Jul-Aug;23(6):412-22. doi: 10.4278/ajhp.080930-QUAN-226. PMID 19601481
- [Background] Zwirska-Korczala K, Konturek SJ, Sodowski M, Wylezol M, Kuka D, Sowa P, Adamczyk-Sowa M, Kukla M, Berdowska A, Rehfeld JF, Bielanski W, Brzozowski T. Basal and postprandial plasma levels of PYY, ghrelin, cholecystokinin, gastrin and insulin in women with moderate and morbid obesity and metabolic syndrome. J Physiol Pharmacol. 2007 Mar;58 Suppl 1:13-35. PMID 17443025
- [Background] Abell TL, Camilleri M, Donohoe K, Hasler WL, Lin HC, Maurer AH, McCallum RW, Nowak T, Nusynowitz ML, Parkman HP, Shreve P, Szarka LA, Snape WJ Jr, Ziessman HA; American Neurogastroenterology and Motility Society and the Society of Nuclear Medicine. Consensus recommendations for gastric emptying scintigraphy: a joint report of the American Neurogastroenterology and Motility Society and the Society of Nuclear Medicine. J Nucl Med Technol. 2008 Mar;36(1):44-54. doi: 10.2967/jnmt.107.048116. Epub 2008 Feb 20. PMID 18287197